CLINICAL TRIAL: NCT05945290
Title: Pre-Analytical Factors Affecting ctDNA Analysis in Early and Locally Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-012665; UH2CA234306 (NIH); U01CA243078 (NIH); NCI-2022-05844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-012665 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Early Stage Breast Carcinoma; Locally Advanced Breast Carcinoma
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (Biospecimen collection, medical record): Patients undergo blood sample collection throughout the study. Patients also undergo collection of leftover tissue samples from SOC procedures and have medical records reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and leftover tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study evaluates pre-analytical factors affecting circulating tumor deoxyribonucleic acid (ctDNA) analysis in breast cancer that not spread beyond the breast and or lymph nodes (early and locally advanced). ctDNA refers to freely circulating tumor DNA fragments found in the blood plasma. Pre-analytical factors such as blood collection tubes, delays in separation of plasma, centrifugation speeds, storage conditions, shipping and DNA extraction methods can all affect ctDNA measurements. Inappropriate processing can cause breaking down of the membrane (lysis) of peripheral blood cells that release background wild-type DNA and may also cause degradation of circulating tumor-specific DNA fragments. Both mechanisms will dilute levels of ctDNA in plasma and make it more difficult to detect. Evaluating the pre-analytical factors of the collection of blood and left over tissue samples for the research of cancer may help researchers to evaluate the impact of the blood collection/processing and long-term storage from patients with locally advanced breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the impact of blood collection/processing. II. To evaluate the impact of long-term storage of plasma and extracted DNA.

OUTLINE: This is an observational study.

Patients undergo blood sample collection throughout the study. Patients also undergo collection of leftover tissue samples from standard of care (SOC) procedures and have medical records reviewed.

ELIGIBILITY:
Inclusion Criteria:

* All women > 18 years of age
* Stage I-III breast cancer
* Subject has consented to IRB 2130-00 Tissue Registry

Exclusion Criteria:

* Stage IV breast cancer
* Unwilling or unable to give consent
* Unable to participate for 1 year
* No one with a concurrent cancer except those diagnosed with an in situ cancer or non-melanoma skin cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-III breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Change in tumor specific circulating tumor deoxyribonucleic acid (ctDNA) levels | Baseline to 5 years
  Will be measured as tumor fraction (%), using TARgeted DIgital Sequencing (TARDIS).

SECONDARY OUTCOMES:
Change in total cell-free DNA concentration | Baseline to 5 years
  Will be measured in genome copies/ml of plasma, using the Quality Assessment (QA) assay.
Change in total cell-free DNA fragment size profile | Baseline to 5 years
  Will be measured as % fragmented, using the Quality Assessment (QA) assay.
Change in tumor-specific circulating tumor deoxyribonucleic acid (ctDNA) fragment size profile | Baseline to 5 years
  Will be measured as average fragment size, using TARgeted DIgital Sequencing (TARDIS).
Background error rate | Baseline to 5 years
  Will be measured as errors per bp sequenced, measured using TARgeted DIgital Sequencing (TARDIS).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Pockaj, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT05945290/ICF_000.pdf